CLINICAL TRIAL: NCT03716050
Title: The Effect of Nitroglycerin Ointment, Fluorescent Angiography, and Incisional Negative Pressure Wound Therapy on Mastectomy Skin Flap Perfusion-Related Problems
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI decision due to slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB00038262
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2019-12-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2019-09

CONDITIONS: Perfusion; Complications
Keywords: breast reconstruction; Breast Cancer; Implant Complication
MeSH Terms: conditions — Breast Neoplasms | interventions — Nitroglycerin; Negative-Pressure Wound Therapy; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 (Other): Breast skin after mastectomy will be clinically examined by the surgeon to determine if there is adequate blood flow to the skin to allow safe coverage of the breast implant. No treatment, including dye study, ointment, or vacuum dressing will be applied to the breast after implant placement.
  Interventions: Other: No treatment
- Group 2 (Active Comparator): Breast skin after mastectomy will be clinically examined by the surgeon, and nitroglycerin (NTG) cream will be applied to the breast skin after implant placement. This cream does not have systemic effects but may improve blood flow to the remnant breast skin after mastectomy.
  Interventions: Drug: Nitroglycerin
- Group 3 (Active Comparator): Breast skin after mastectomy will be clinically examined by the surgeon, and an incisional vacuum-assisted dressing (iVAC) will be placed over the breast incisions after implant placement, which may improve blood flow to the skin and help wound healing.
  Interventions: Device: Negative Pressure Wound Therapy/ Wound VAC
- Group 4 (Active Comparator): Breast skin after mastectomy will be clinically examined by the surgeon, and both NTG cream will be applied to the breast skin and an iVAC will be placed over the incisions after implant placement.
  Interventions: Drug: Nitroglycerin; Device: Negative Pressure Wound Therapy/ Wound VAC
- Group 5 (Active Comparator): Blood flow to breast skin after mastectomy will be examined using a fluorescent dye study called fluorescent angiography (FA) to determine if there is adequate blood flow to the skin to allow safe coverage of the breast implant. No further intervention will be used after implant placement.
  Interventions: Other: Fluorescent Angiography with indocyanine-green (not to exceed 5mg/kg)
- Group 6 (Active Comparator): Blood flow to breast skin breast skin will be examined using FA, and NTG cream will be applied to the skin after the implant is placed.
  Interventions: Drug: Nitroglycerin; Other: Fluorescent Angiography with indocyanine-green (not to exceed 5mg/kg)
- Group 7 (Active Comparator): Blood flow to breast skin breast skin will be examined using FA, and an iVAC will be placed over breast skin incisions after the implant is placed.
  Interventions: Device: Negative Pressure Wound Therapy/ Wound VAC; Other: Fluorescent Angiography with indocyanine-green (not to exceed 5mg/kg)
- Group 8 (Active Comparator): Blood flow to breast skin breast skin will be examined using FA, and both NTG cream and iVAC will be used as interventions after the implant is placed.
  Interventions: Drug: Nitroglycerin; Device: Negative Pressure Wound Therapy/ Wound VAC; Other: Fluorescent Angiography with indocyanine-green (not to exceed 5mg/kg)

INTERVENTIONS:
Drug: Nitroglycerin — Patient's will be randomized into one of eight groups and receive the intended treatment specified for that particular group. Groups 2,4,6, and 8 will include Nitroglycerin cream.
  Other Names: Nitro-Bid 2%
  Arms: Group 2; Group 4; Group 6; Group 8
Device: Negative Pressure Wound Therapy/ Wound VAC — Patient's will be randomized into one of eight groups and receive the intended treatment specified for that particular group. Groups 3,4,7,and 8 will receive iVAC therapy.
  Other Names: iVAC
  Arms: Group 3; Group 4; Group 7; Group 8
Other: Fluorescent Angiography with indocyanine-green (not to exceed 5mg/kg) — Patient's will be randomized into one of eight groups and receive the intended treatment specified for that particular group. Groups 5,6,7,and 8 will receive angiography.
  Arms: Group 5; Group 6; Group 7; Group 8
Other: No treatment — Patient's will be randomized into one of eight groups and receive the intended treatment specified for that particular group. Groups 1 will include no treatment.
  Arms: Group 1

SUMMARY:
This is a randomized study using a variety of techniques to compare and examine blood flow to the remaining skin after mastectomy. All treatments being used are considered standard of care and are not experimental. The objective is to compare the techniques and the incidence of perfusion related problems in patient's undergoing mastectomy with immediate breast reconstruction.

DETAILED DESCRIPTION:
This study's aim is to evaluate and compare a variety of interventions and their effect on the incidence of perfusion related problems in patients with breast cancer undergoing mastectomy and implant-based immediate breast reconstruction (IBR). The ability to identify, prevent and treat these perfusion related problems can help maximize aesthetic results after breast surgery, improve patient satisfaction with both mastectomy and breast reconstruction, and reduce healthcare cost associated with mastectomy and reconstruction complications.The study team will perform a randomized pilot study comprised of eight groups. All of these groups employ accepted techniques, medications and dressings and therefore are not experimental.

Group 1: Breast skin after mastectomy will be clinically examined by the surgeon to determine if there is adequate blood flow to the skin to allow safe coverage of the breast implant. No dye study, ointment, or vacuum dressing will be applied to the breast after implant placement.

Group 2 - Breast skin after mastectomy will be clinically examined by the surgeon, and nitroglycerin (NTG) cream will be applied to the breast skin after implant placement. This cream does not have systemic effects but may improve blood flow to the remnant breast skin after mastectomy.

Group 3 - Breast skin after mastectomy will be clinically examined by the surgeon, and an incisional vacuum-assisted dressing (iVAC) will be placed over the breast incisions after implant placement, which may improve blood flow to the skin and help wound healing.

Group 4 - Breast skin after mastectomy will be clinically examined by the surgeon, and both NTG cream will be applied to the breast skin and an iVAC will be placed over the incisions after implant placement.

Group 5 - Blood flow to breast skin after mastectomy will be examined using a fluorescent dye study called fluorescent angiography (FA) to determine if there is adequate blood flow to the skin to allow safe coverage of the breast implant. No further intervention will be used after implant placement.

Group 6 - Blood flow to breast skin breast skin will be examined using FA, and NTG cream will be applied to the skin after the implant is placed.

Group 7 - Blood flow to breast skin breast skin will be examined using FA, and an iVAC will be placed over breast skin incisions after the implant is placed.

Group 8 - Blood flow to breast skin breast skin will be examined using FA, and both NTG cream and iVAC will be used as interventions after the implant is placed.

The dosage of indocyanine-green (IC-green) to be used for assessment of mastectomy flaps will be in 10 mg boluses, not to exceed 5 mg/kg.

Nitro-Bid® (nitroglycerin ointment, 2%) at a dose of 45 mg (equal to 7.5 cm on the measuring strip provided with packaging) will be used. The paste will be applied to remnant breast skin after skin closure and surgical dressings placed over top.

Incisional negative pressure wound therapy will consist of a standard sponge dressing with adhesive drape, either Ioban® 2 (3M ™) or KCI-V.A.C.® Drape (KCI®), to continuous suction at 125 mm Hg while the patient is in hospital and not to exceed 4 days.

A physician will see the subjects on a regular weekly basis for up to 30 days once the procedure has been completed. These clinical visits are standard of care and the subject's health and well-being will be monitored rigorously during these visits. If during any of these visits, the physician deems a therapy necessary to prevent impairment/damage and improve well-being, the subject will be treated appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female.
* Patients must be between the ages of 18 and 99 years.
* Patients must undergo mastectomy with our attending breast oncology surgeons followed by possible implant-based immediate breast reconstruction (IBR) performed by our attending plastic surgeons at WFBMC.
* Patients must have the ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Patients who are under the age of 18 or over the age of 99.
* Patients who are undergoing mastectomy without immediate breast reconstruction including immediate breast reconstruction with autologous tissue (or combination of autologous tissue with tissue expanders or implants), or patients with a history of mastectomy presenting for delayed breast reconstruction.
* Patients with pre-existing conditions in which use of indocyanine-green is contraindicated or must be used with caution, including those with a history of allergy to iodides or iodinated dye, those with chronic kidney disease, those with hepatic failure or cirrhosis of the liver, and females who are nursing, pregnant, or may become pregnant.
* Pregnant women are excluded from this study because pregnancy precludes immediate breast reconstruction in our patient population.
* Patients with pre-existing conditions in which use of nitroglycerin paste is contraindicated, including those with a history of cardiac insufficiency, hypotension, sensitivity to nitrites, severe liver impairment, glaucoma, hyperthyroidism, recent head trauma, severe anemia, or taking certain medication (i.e. alteplase, aspirin, beta-blocker, calcium channel blocker, diuretics or thiazides).
* Patients with pre-existing conditions in whom use of incisional negative pressure wound therapy is contraindicated including those with evidence of surgical site infection ( i.e. erythema, purulent drainage), clinical signs of hematoma (i.e. wound swelling, fluctuance, blood drainage), history of persistent cancer, exposed blood vessel on site of proposed therapeutic use, or sensitivity to acrylics and adhesives.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient's must be females, diagnosed with breast cancer and desiring breast reconstruction
Enrollment: 17 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivo A Pestana, MD, Principal Investigator — WFUHS
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8
Started | 2 | 4 | 1 | 3 | 1 | 0 | 4 | 2
Completed | 2 | 4 | 0 | 1 | 1 | 0 | 4 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: There were no participants randomized to group 6
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Total
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 0 | 4 | 2 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 2 | 0 | 0 | 4 | 2 | 14
  >=65 years | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 3 | 1 | 0 | 4 | 2 | 17
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 1 | 3 | 1 | 0 | 4 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Soft Tissue Ischemia/Loss
Description: Number of partial and full thickness soft tissue defects identified postoperatively in clinic follow up
Time Frame: Up to 30 days
Population: There were no participants randomized to group 6
Measure: Number; unit: number of defects
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
number of defects | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Surgical Site Infection
Description: Number of Participants with soft tissue cellulitis or abscess identified postoperatively either clinically or with wound culture
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Delayed Wound Healing
Description: manifesting as suture dehiscence and opening of an incisional wound
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Operative Intervention Secondary to Perfusion Related Problems
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Requiring Outpatient Prescription for Antibiotics or Requiring Hospital Admission for IV Antibiotics
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Requiring Wound Care Management Modalities for Treatment of Delayed Wound Healing Complications
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 7 | Group 8
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 1 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time subjects sign consent through Week 4 (30 days)
Description: There were no subjects randomized to group 6
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/1 | 0/3 | 0/1 | 0/0 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/1 | 0/3 | 0/1 | 0/0 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/1 | 0/3 | 0/1 | 0/0 | 1/4 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=2) | Group 2 (N=4) | Group 3 (N=1) | Group 4 (N=3) | Group 5 (N=1) | Group 6 (N=0) | Group 7 (N=4) | Group 8 (N=2)
Pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain with removal of wound VAC

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03716050/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03716050/ICF_001.pdf